Mindfulness + tDCS to reduce urgency incontinence in women

NCT# 04652869

Study Protocol 9/13/2022

## Scientific background

Urinary incontinence, particularly urinary urge incontinence (UUI), is a highly prevalent and costly (\$83 billion/year) disorder among older women. Greater than 50% of UUI-related urgency and leakage may be due to situational incontinence provoked by confrontation with specific contextual triggers or cues (e.g., seeing one's front/garage door, doing dishes). We recently found that women with UUI experience increased urgency and actual leakage when exposed to personal "urge" versus "safe" photographic cues taken from their daily lives. Decades of cuebased research across other disorders has shown that such conditioned responses are rarely attenuated with pharmacologic methods and require cognitive and behavioral retraining. Therefore, new methods are needed to specifically target conditioned factors contributing to UUI, in order to effectively combat this persistent contributor to urgency and leakage and augment the efficacy of current UUI treatments.

We propose to test two new intervention methods to attenuate UUI symptomatology and reactivity to urgency cues among women with situational UUI. These methods include brief mindfulness (MI) and transcranial direct current stimulation (tDCS). Employing our well-tested method to personalize cues, women with situational UUI will create photographic personal "urge" cues, which capture their strongest urgency, and "safe" cues, in which they do not experience urge. Then, we will examine the feasibility, acceptability, participant compliance, and efficacy of using MI and/or tDCS to reduce cue-provoked urgency and/or leakage to these salient personal cues, reduce reaction time on a urinary Stroop test, and decrease multiple UUI outcomes.

## **Study Objectives:**

Aim 1: Assess intervention feasibility, acceptability, and compliance. <u>H1: Feasibility:</u> 85% of all enrolled participants will complete the study, <u>Acceptability:</u> Moderate to high acceptability rating of  $\geq$  50 (0-100 scale) and <u>Participant compliance:</u>  $\geq$  75 (0-100 scale) for MI compliance on the self-reported post-study survey.

**Aim 2: Examine UUI symptom reduction**. <u>H1:</u> Each intervention will lead to a pre-post and pre-follow-up reduction in number of UUI episodes, self-report urgency, and bladder symptom severity (ICIQ-FLUTS). <u>H2:</u> MI + tDCS will lead to the greatest reduction in these UUI symptoms.

Aim 3: Examine attenuation of reactivity to urgency stimuli. <u>H1</u>: Each intervention will reduce cue-reactivity and urinary Stroop reaction time. <u>H2</u>: MI + tDCS will lead to greater reductions in these measures relative to either MI or tDCS alone.

## Study Design and methods

We will examine the independent and combined effects of brief mindfulness (MI) and transcranial direct current stimulation (tDCS) across three group: 1) MI, 2) tDCS, 3) MI + tDCS. MI and / or tDCS will be employed during urgency-cue exposure to examine the efficacy of these methods to attenuate cue reactivity (cue-induced urgency, reaction time during a urinary Stroop test) and lead to reductions in self-reported bladder problem severity (ICIQ-FLUTS score), UUI episodes, and urgency ratings. Some participants will be trained in a brief mindfulness intervention (MI; 20-minute audio guide) to focus on body scan with acceptance language and will practice it out of session to use during cue exposure. Second, transcranial direct current stimulation (tDCS) targeting the dorsolateral prefrontal cortex (dIPFC) with be used to increase cortical excitability in the dIPFC, aimed at increasing cognitive control when confronted with personal urgency cues. tDCS has been shown to reduce cue reactivity on its own, and we will also test it as such, but research has also shown augmentation of its effectiveness when paired with tasks that engage brain regions being targeted for related behavior change. Past research has shown that mindfulness engages the PFC and that women with UUI who are not responsive to pharmacotherapy demonstrate down regulation of the PFC,

suggesting that tDCS combined with MI should further enhance cognitive control over reactivity to cue-provoked urgency and reduce UUI-related outcomes.

#### **Procedures and Protocols**

Sixty women will be recruited from the Pitt+Me online registry, local fliers and through collaboration with multiple community and university resources (see recruitment). Telephone screening will determine initial eligibility. Eligible participants will be invited to Dr. Conklin's laboratory for informed consent, further screening, and a semi-structured interview to identify personal urgency and safe cue environments, of which each participant will take pictures. Participants will then be randomized to one of 3 groups: 1) Mindfulness, 2) tDCS, 3) Mindfulness + tDCS. We will use the SAS® high quality pseudorandom deviate generator (SAS Institute, Cary, NC) to randomize subjects in a 1:1:1 ratio. We will use a blocked randomization scheme to force an approximate balance between the number of subjects in each arm at any point during recruitment. Participants will undergo 4 urgency cue exposure sessions with their assigned intervention. Cue-induced urgency and reaction time to modified Stroop will be assessed at baseline and post-training. Bladder diary and urgency survey will be completed daily throughout the study, and for one-week post-training.

#### Interventions:

1) Brief Mindfulness (Body Scan with awareness/acceptance language): Imaging studies have revealed enhanced activation of the PFC<sup>1</sup>, and more specifically the dIPFC<sup>2,3</sup>, during mindfulness practice, and while completing executive processing tasks after MI training. During mindfulness training, practitioners cultivate a nonjudgmental state of attention to experiences in the present moment4, resulting in active engagement of attentional control abilities<sup>5-7</sup>. Recent work on MI-based stress reduction (MBSR) to attenuate UUI symptoms found significant reductions in UUI episodes post-treatment, with continued reduction over 6 months post-treatment, suggesting increased benefit over time<sup>8,9</sup>. Mindfulness has also been shown to reduce cue reactivity, with significant reductions in cue responding to food<sup>10</sup>, anxiety<sup>11</sup>, addiction <sup>12-14</sup>, and mood regulation <sup>15</sup> cues following MI training, presumed to reflect increased cognitive control over salient disorder-related stimuli. Recently, less intensive brief mindfulness interventions (i.e., significantly less than 8-week MBSR) have been tested with positive results. 16-20 This work has shown immediate beneficial effects on anxiety 18, coping with social stressors<sup>3</sup>, acute pain<sup>20</sup> and increasing self-control,<sup>19</sup> without requiring a full MBSR program<sup>21</sup>. Brief interventions are lower cost, less burdensome and more accessible at home, which is attractive for a self-management care model for chronic illness.<sup>22,23</sup> Given the success in reducing UUI episodes following the full 8-week MBSR program<sup>8,9</sup> UUI is a particularly good candidate for testing new brief mindfulness methods.

A component of MBSR commonly isolated for brief intervention is body scan<sup>24</sup>. This method involves focused attention on the present moment through observing one's breath and bodily sensations, while becoming aware of, and accepting without judgement, any thoughts and feelings that arise.<sup>25</sup> Body scans are used for brief mindfulness training in both clinical and research protocols, and typically last between 5 and 30 min<sup>20,21</sup>. We will test a novel MI presented and practiced with a 15-minute guided audio recording consisting of guidance to attend to physical sensations with a gentle, accepting attitude.

<u>2) Transcranial Direct Current Stimulation (tDCS)</u>: tDCS is a safe, non-invasive method of brain stimulation that **can enhance cortical excitability and help attenuate cue-induced reactivity**. tDCS has become increasingly popular in clinical and neurocognitive research, showing promising efficacy for targeting cue-reactivity to stimuli related to a number of disorders (depression, addiction, anxiety), assisting physical and cognitive recovery secondary to stroke and spinal cord injury<sup>26-28</sup>, and promoting cognitive enhancement in healthy subjects.<sup>29-</sup>

<sup>32</sup> Addiction research incorporating tDCS has shown reductions in cue-induced craving in response to drug-related stimuli from baseline to re-test following a single session of tDCS,<sup>33</sup> as well as reductions in cue-induced craving and actual smoking after 3-5 tDCS sessions.<sup>34</sup>

In anxiety research, reductions in self-reported and physiological reactivity to fear stimuli have been noted after similar tDCS methods<sup>35</sup>. These effects have been characterized through consideration of the PFC's role in decision-making and cognitive control and are presumed to reflect increased control over cue reactivity following PFC-targeted tDCS. Although effective as a standalone treatment to reduce reactivity, the effects of tDCS are greatly enhanced when stimulation is paired with behavioral training that engages the brain processes that underlie the targeted behavior.<sup>36</sup> Thus, we purport that brief mindfulness during urgency-cue exposure is a prime candidate for augmentation with dIPFC-targeted tDCS. Enhancement of excitability in the PFC during mindfulness, which has also been shown to increase dIPFC activation<sup>3,37,38</sup> and cognitive control<sup>39</sup> should lead to greater ability to dynamically recruit cognitive control systems during urgency situations, which will aid in retraining the salience of urgency-related cues.

# **Inclusion Criteria:**

- Ambulatory women aged 40+ years
- Able to differentiate between stress symptoms (cough, laugh, exercise) and urgency symptoms (leakage following sudden strong urge to void that is difficult to defer), and history suggestive of UUI using our detailed incontinence history questionnaires and clinical expertise.
- self-report of 2 leaks/week,
- Self-report of 'sometimes' or 'often' experiencing urgency or leakage in at least 4 of 15 common urgency trigger scenarios
- A bother score ≥4 on a situational urgency questionnaire
- Subjects using OAB medication will be considered if they have used it consistently for 3 months and plan to keep using it throughout the duration of the study.

## **Exclusion criteria:**

- Inability to reliably describe incontinence type (i.e. Inability to identify situational urgency trigger scenarios, differentiate between stress and urgency incontinence, describe leakage scenarios.)
- Cognitive impairment (inability to: accurately complete a bladder diary, identify and take appropriate photos of urge cue and safe cue scenarios, appropriately give incontinence history)
- Spinal cord injury; history of pelvic irradiation, advanced uterine or bladder cancer
- Urinary retention [PVR >200 ml]
- Interstitial cystitis; artificial sphincter implant
- Medical instability or expected change in medication during the study (e.g. change in anticholinergic, diuretic medication)
- Conditions that preclude tDCS including: Epilepsy or current seizure disorder, pregnant or lactating, implanted cardiac or brain medical device.

**Primary Outcomes: Data Analysis Plan.** Prior to hypothesis testing, descriptive statistics and graphic displays will be used to identify outliers, missing data, and patterns of attrition, and to guide transformations and appropriate tests. The primary analyses will be evaluated via mixed model regressions with Bonferroni post-hoc comparisons. Mixed model regression features advantages over traditional regression due to the ability to handle repeated assessments of both predictor variables and outcome variables. For **Aim 1**, We will assess feasibility as >85% study

completion, acceptability as a score ≥50 on 8-item post-study survey rating (scale 0-100), and mindfulness compliance as an average rating ≥75 on the compliance survey (scale 0-100). We will use chi-square to assess attrition differences between groups, and one-way ANOVA to assess differences in acceptability and compliance ratings. For <u>Aim 2</u>, mixed model regressions will test the main effects of experimental group (1=MI, 2=tDCS, and 3=MI+tDCS) on ICIQ-FLUTS score (pre, post, and follow-up), UUI episodes, and urgency survey scores (3-day mean score at baseline, last three days before re-test, and last 3-days of follow-up) as dependent variables. Pre-intervention (baseline) levels of each dependent variable will be entered as a covariate in respective regression models. This process will be repeated for <u>Aim 3</u>, with separate models evaluating treatment effects on Stroop RT and cue-provoked urgency. For Stroop RT, the primary dependent variable will be post-test minus pre-test change. For cue-provoked urgency, the primary dependent variable will represent a double-difference score of urgency minus safe cues, and post-test minus test.

- 1. Chiesa A, Serretti A. A systematic review of neurobiological and clinical features of mindfulness meditations. Psychological Medicine. 2010;40(8):1239-52. doi: 10.1017/S0033291709991747.
- 2. Allen M, Dietz M, Blair KS, van Beek M, Rees G, Vestergaard-Poulsen P, Lutz A, Roepstorff A. Cognitive-affective neural plasticity following active-controlled mindfulness intervention. Journal of Neuroscience. 2012;32(44):15601–10.
- 3. Creswell JD, Pacilio LE, Lindsay EK, Brown KW. Brief mindfulness meditation training alters psychological and neuroendocrine responses to social evaluative stress. Psychoneuroendocrinology. 2014;44:1-12. doi: 10.1016/j.psyneuen.2014.02.007.
- 4. Kabat-Zinn J, Lipworth L, Burney R. The clinical use of mindfulness meditation for the self-regulation of chronic pain. Journal of behavioral medicine. 1985;8(2):163–90.
- 5. Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. Journal of personality and social psychology. 2003;84(4):822.
- 6. Lutz A, Slagter HA, Dunne JD, Davidson RJ. Attention regulation and monitoring in meditation. Trends Cogn Sci. 2008;12(4):163–9.
- 7. Malinowski P. Neural mechanisms of attentional control in mindfulness meditation. Frontiers in neuroscience. 2013;7:8.
- 8. Baker J, Costa D, Nygaard I. Mindfulness-Based Stress Reduction for Treatment of Urinary Urge Incontinence: A Pilot Study. Female Pelvic Medicine & Reconstructive Surgery. 2012;18(1):46. doi: 10.1097/SPV.0b013e31824107a6.
- 9. Baker J, Costa D, Guarino JM, Nygaard I. Comparison of Mindfulness-Based Stress Reduction Versus Yoga on Urinary Urge Incontinence: A Randomized Pilot Study. With 6-Month and 1-Year Follow-up Visits. Female Pelvic Medicine & Reconstructive Surgery. 2014;20(3):141. doi: 10.1097/SPV.000000000000001.
- 10. Keesman M, Aarts H, Häfner M, Papies EK. Mindfulness Reduces Reactivity to Food Cues: Underlying Mechanisms and Applications in Daily Life. Current Addiction Reports. 2017;4(2):151-7. doi: 10.1007/s40429-017-0134-2.
- 11. Hofmann SG, Sawyer AT, Witt AA, Oh D. The effect of mindfulness-based therapy on anxiety and depression: A meta-analytic review. Journal of Consulting and Clinical Psychology. 2010;78(2):169-83. doi: 10.1037/a0018555.
- 12. Garland EL. Trait Mindfulness Predicts Attentional and Autonomic Regulation of Alcohol Cue-Reactivity. J Psychophysiol. 2011;25(4):180-9. doi: 10.1027/0269-8803/a000060. PubMed PMID: 23976814.

- 13. Garland EL, Froeliger B, Howard MO. Effects of Mindfulness-Oriented Recovery Enhancement on reward responsiveness and opioid cue-reactivity. Psychopharmacology. 2014;231(16):3229-38. Epub 03/05. doi: 10.1007/s00213-014-3504-7. PubMed PMID: 24595503.
- 14. Janes AC, Datko M, Roy A, Barton B, Druker S, Neal C, Ohashi K, Benoit H, van Lutterveld R, Brewer JA. Quitting starts in the brain: a randomized controlled trial of app-based mindfulness shows decreases in neural responses to smoking cues that predict reductions in smoking. Neuropsychopharmacology. 2019. doi: 10.1038/s41386-019-0403-y.
- 15. Guendelman S, Medeiros S, Rampes H. Mindfulness and Emotion Regulation: Insights from Neurobiological, Psychological, and Clinical Studies. Frontiers in psychology. 2017;8:220-. doi: 10.3389/fpsyg.2017.00220. PubMed PMID: 28321194.
- 16. Bergen-Cico D, Possemato K, Cheon S. Examining the efficacy of a brief mindfulness-based stress reduction (brief MBSR) program on psychological health. Journal of American College Health. 2013;61(6):348–60.
- 17. Bowen S, Marlatt A. Surfing the urge: Brief mindfulness-based intervention for college student smokers. Psychology of Addictive Behaviors. 2009;23(4):666-71. doi: 10.1037/a0017127.
- 18. Call D, Miron L, Orcutt H. Effectiveness of brief mindfulness techniques in reducing symptoms of anxiety and stress. Mindfulness. 2014;5(6):658–68.
- 19. Canby NK, Cameron IM, Calhoun AT, Buchanan GM. A brief mindfulness intervention for healthy college students and its effects on psychological distress, self-control, meta-mood, and subjective vitality. Mindfulness. 2015;6(5):1071–81.
- 20. Zeidan F, Gordon NS, Merchant J, Goolkasian P. The Effects of Brief Mindfulness Meditation Training on Experimentally Induced Pain. The Journal of Pain. 2010;11(3):199-209. doi: 10.1016/j.jpain.2009.07.015.
- 21. Zeidan F, Johnson SK, Diamond BJ, David Z, Goolkasian P. Mindfulness meditation improves cognition: Evidence of brief mental training. Consciousness and cognition. 2010;19(2):597–605.
- 22. Bodenheimer T, Lorig K, Holman H, Grumbach K. Patient self-management of chronic disease in primary care. Jama. 2002;288(19):2469–75.
- 23. Von Korff M, Gruman J, Schaefer J, Curry SJ, Wagner EH. Collaborative management of chronic illness. Annals of internal medicine. 1997;127(12):1097–102.
- 24. Cropley M, Ussher M, Charitou E. Acute effects of a guided relaxation routine (body scan) on tobacco withdrawal symptoms and cravings in abstinent smokers. Addiction. 2007;102(6):989-93. doi: 10.1111/j.1360-0443.2007.01832.x.
- 25. Witkiewitz K KMFTAMLMERCOSAJBDHMCBA, Clark VP. Mindfulness and Transcranial Direct Current Stimulation as an Intervention for Tobacco Dependence: A Pilot Study2015.
- 26. Schlaug G, Renga V, Nair D. Transcranial Direct Current Stimulation in Stroke Recovery. Archives of neurology. 2008;65(12):1571-6. doi: 10.1001/archneur.65.12.1571. PubMed PMID: PMC2779259.
- 27. Cortes M, Medeiros AH, Gandhi A, Lee P, Krebs HI, Thickbroom G, Edwards D. Improved grasp function with transcranial direct current stimulation in chronic spinal cord injury. NeuroRehabilitation. 2017;41(1):51-9. Epub 2017/05/17. doi: 10.3233/nre-171456. PubMed PMID: 28505987.
- 28. Gunduz A, Rothwell J, Vidal J, Kumru H. Non-invasive brain stimulation to promote motor and functional recovery following spinal cord injury. Neural regeneration research. 2017;12(12):1933-8. Epub 2018/01/13. doi: 10.4103/1673-5374.221143. PubMed PMID: 29323025; PMCID: PMC5784334.
- 29. Clark VP, Coffman BA, Mayer AR, Weisend MP, Lane TDR, Calhoun VD, Raybourn EM, Garcia CM, Wassermann EM. TDCS guided using fMRI significantly accelerates learning to identify concealed objects. NeuroImage. 2012;59(1):117–28.
- 30. Falcone B, Coffman BA, Clark VP, Parasuraman R. Transcranial direct current stimulation augments perceptual sensitivity and 24-hour retention in a complex threat detection task. PLoS ONE. 2012;7(4):e34993.

- 31. Marshall L, Mölle M, Hallschmid M, Born J. Transcranial direct current stimulation during sleep improves declarative memory. The Journal of neuroscience. 2004;24(44):9985–92.
- 32. Ragert P, Vandermeeren Y, Camus M, Cohen LG. Improvement of spatial tactile acuity by transcranial direct current stimulation. Clinical Neurophysiology. 2008;119(4):805–11.
- 33. Fregni F, Liguori P, Fecteau S, Nitsche MA, Pascual-Leone A, Boggio PS. Cortical stimulation of the prefrontal cortex with transcranial direct current stimulation reduces cue-provoked smoking craving: a randomized, sham-controlled study. Journal of Clinical Psychiatry. 2008;69(1):32–40.
- 34. Boggio PS, Liguori P, Sultani N, Rezende L, Fecteau S, Fregni F. Cumulative priming effects of cortical stimulation on smoking cue-induced craving. Neurosci Lett. 2009;463(1):82-6. doi: 10.1016/j.neulet.2009.07.041.
- 35. Dittert N, Hüttner S, Polak T, Herrmann MJ. Augmentation of Fear Extinction by Transcranial Direct Current Stimulation (tDCS). Front Behav Neurosci. 2018;12. doi: 10.3389/fnbeh.2018.00076.
- 36. Gill J, Shah-Basak PP, Hamilton R. It's the thought that counts: examining the task-dependent effects of transcranial direct current stimulation on executive function. Brain Stimulation: Basic, Translational, and Clinical Research in Neuromodulation. 2015;8(2):253–9.
- 37. Creswell JD, Taren AA, Lindsay EK, Greco CM, Gianaros PJ, Fairgrieve A, Marsland AL, Brown KW, Way BM, Rosen RK, Ferris JL. Alterations in Resting-State Functional Connectivity Link Mindfulness Meditation With Reduced Interleukin-6: A Randomized Controlled Trial. Biol Psychiatry. 2016;80(1):53-61. Epub 2016/03/30. doi: 10.1016/j.biopsych.2016.01.008. PubMed PMID: 27021514.
- 38. Taren AA, Gianaros PJ, Greco CM, Lindsay EK, Fairgrieve A, Brown KW, Rosen RK, Ferris JL, Julson E, Marsland AL, Bursley JK, Ramsburg J, Creswell JD. Mindfulness meditation training alters stress-related amygdala resting state functional connectivity: a randomized controlled trial. Soc Cogn Affect Neurosci. 2015;10(12):1758-68. Epub 2015/06/07. doi: 10.1093/scan/nsv066. PubMed PMID: 26048176; PMCID: PMC4666115.
- 39. Hunter MA, Lieberman G, Coffman BA, Trumbo MC, Armenta ML, Robinson CSH, Bezdek MA, O'Sickey AJ, Jones AP, Romero V, Elkin-Frankston S, Gaurino S, Eusebi L, Schumacher EH, Witkiewitz K, Clark VP. Mindfulness-based training with transcranial direct current stimulation modulates neuronal resource allocation in working memory: A randomized pilot study with a nonequivalent control group. Heliyon. 2018;4(7):e00685. doi: 10.1016/j.heliyon.2018.e00685. PubMed PMID: PMC6077241.